CLINICAL TRIAL: NCT04844567
Title: Virtual Reality Intervention Alleviates Dyspnea in Patients Recovering From COVID Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Collaborators: Mindmaze SA (Industry)
Responsible Party: Principal Investigator, Olaf Blanke, Professor Doctor, Ecole Polytechnique Fédérale de Lausanne
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: COVVR_LNCO2020
Record Dates: First submitted 2021-03-18; First posted 2021-04-14 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Covid19; Dyspnea
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Intervention Model Description: Participants perform both conditions. Condition order was randomised across participants using a script prior to data collection.
Who Masked: Participant, Care Provider
Masking Description: Participants are naïve to the difference in interventions. Allocation was concealed to the care provider screening participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVVR_A (Experimental): Participants in the COVVR_A arm complete the synchronous block first, followed by the asynchronous block.
  Interventions: Device: COVVR_Synch; Device: COVVR_Asynch
- COVVR_B (Experimental): Participants in the COVVR_B arm complete the asynchronous block first, followed by the synchronous block.
  Interventions: Device: COVVR_Synch; Device: COVVR_Asynch

INTERVENTIONS:
Device: COVVR_Synch — Participants wear a respiration belt (Vernier, Go Direct) that continuously transmits thoracic circumference readings to a mobile phone (Samsung Galaxy S8) in real-time. The mobile device is placed in a headset (Zeiss VR ONEPLUS) and used to create a stereoscopic, immersive scene in Virtual Reality. The data from the respiration belt is used to map the on-going respiration pattern onto a virtual body in the scene in one of two feedback conditions.
  COVVR_Synch provided synchronous feedback: participants receive real-time feedback of their respiration.
Device: COVVR_Asynch — Participants wear a respiration belt (Vernier, Go Direct) that continuously transmits thoracic circumference readings to a mobile phone (Samsung Galaxy S8) in real-time. The mobile device is placed in a headset (Zeiss VR ONEPLUS) and used to create a stereoscopic, immersive scene in Virtual Reality. The data from the respiration belt is used to map the on-going respiration pattern onto a virtual body in the scene in one of two feedback conditions.
  COVVR_Asynch provided asynchronous feedback: participants receive asynchronous, frequency modulated feedback of their respiration.

SUMMARY:
The present COVID-19 Virtual Reality (COVVR) clinical study is performed to test the hypothesis that an immersive virtual reality (iVR)-based Digital Therapeutics (DTx), would alleviate dyspnea by improving breathing comfort in patients recovering from COVID-19 pneumonia presenting with persistent dyspnea. We will further evaluate participants' perceived awareness of and agency over their breathing movements. Finally, we will track patients' perceived benefits related to the iVR intervention and the feasibility of using COVVR in the clinic or at home.

DETAILED DESCRIPTION:
Persistent dyspnea is the experience of breathlessness that persists despite optimal treatment of the underlying pathophysiology, and results in physical, psychosocial disability for the patient. As observed for SARS-CoV and MERS-CoV patients, a significant portion of COVID-19 patients present with persistent respiratory physiological impairment and persistent breathlessness that may not be addressed with conventional respiratory treatment such as oxygen, bronchodilators, diuretics or non-invasive ventilation.

Previous research on respiration-related feedback in Virtual Reality (VR) has demonstrated strong and replicable effects of VR feedback over one's perceived sense of agency and control over one's virtually embodied respiration. Based on these studies, the VR intervention evaluated here aims to alleviate symptoms of perceived breathlessness.

This within-subject study will compare breathing comfort as well as breathing discomfort, prior, during, and after a VR intervention that provides embodied visual feedback of participants' on-going respiration. Primary outcomes include subjective reports from participants (breathing comfort and breathing discomfort) and the intervention's clinical feasibility. Secondary outcomes include subjective ratings on perceived embodiment and sense of agency, as well as changes in respiration rate and variability.

ELIGIBILITY:
Inclusion Criteria:

* Recovering from COVID-19 pneumonia confirmed by RT-PCR for SARS-CoV-2
* Presented with persistent dyspnea with a self-rated intensity of five or higher (out of ten) on a visual analog dyspnea scale. ( "Do you have difficulty breathing?" "On a scale of 0 to 10, with 0 being no difficulty to breathe and 10 being the worst difficulty to breathe that you can imagine, where do you rank?".) This dyspnea rating will only used as an inclusion criterion and not as an outcome.
* Being able to give consent
* Being able to understand and speak French or English

Exclusion Criteria:

* Any unstable respiratory, neurological, and cardiac conditions
* Any psychiatric illness
* Montreal Cognitive Assessment (MoCA) score below 25.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Efficacy (Breathing Comfort & Discomfort) | through study completion, an average of one year
  Efficacy will be evaluated based on subjective feedback by the patients regarding their breathing comfort and discomfort, depending on the intervention.
  Subjective ratings will be measured using a 7-point Likert scale with -3 = Strongly disagree, -2 = Disagree; -1 = Somewhat disagree; 0 = Neither agree nor disagree; 1 = Somewhat agree; 2 = Agree; 3= Strongly agree.
  Comfort item: "My breathing was enjoyable" Discomfort item: "I had difficulty breathing"
VR Intervention Feasibility | through study completion, an average of one year
  Feasibility will be evaluated using a feedback questionnaire, alongside open feedback. Agreement with the questionnaire items indicates better feasibility, acceptance, and perceived outcome.
  Ratings will be measured using a 7-point Likert scale with -3 = Strongly disagree, -2 = Disagree; -1 = Somewhat disagree; 0 = Neither agree nor disagree; 1 = Somewhat agree; 2 = Agree; 3= Strongly agree.
  Satisfaction: Did you enjoy the VR experience? Rehabilitation: Would you like to continue using the device during your recovery? Hospital Use: Would you have liked to use this earlier during your stay at the hospital? Home Use: Would you like to continue using the device at home? Respiratory benefit: Do you think the VR feedback improved your breathing? Well-being benefit: Did the VR feedback make you feel better?

SECONDARY OUTCOMES:
Embodiment | through study completion, an average of one year
  Change in subjective ratings about embodiment depending on VR intervention. Two control items are included that are not expected to change between conditions.
  Ratings will be measured using a 7-point Likert scale with -3 = Strongly disagree, -2 = Disagree; -1 = Somewhat disagree; 0 = Neither agree nor disagree; 1 = Somewhat agree; 2 = Agree; 3= Strongly agree.
  Breathing awareness: It seemed as if the flashing was my respiration Control 1: It seemed as if I had three bodies Breathing agency: I felt as if the virtual body was breathing with me Control 2: I felt as if the virtual body was drifting with the flashing
Respiratory Rate | through study completion, an average of one year
  Change in respiratory rate depending on VR intervention. Respiratory rate (RR) will be measured in breaths per minute. RR will be assessed with respect to baseline recordings.
Respiratory Rate Variability | through study completion, an average of one year
  Change in respiratory rate variability depending on VR intervention. Respiratory rate variability (RRV) will be measured using inter-breath intervals (IBI).
  RRV will be assessed with respect to baseline recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Blanke, Prof, Principal Investigator — Ecole Polytechnique Fédérale de Lausanne
Locations (1):
- Hopitaux Universitaires de Geneve (HUG), Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No